CLINICAL TRIAL: NCT00050804
Title: Efficacy of an SSRI in Acute Stress Disorder and PTSD
Brief Title: Evaluation of Stress Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 030036; 03-M-0036
Record Dates: First submitted 2002-12-19; First posted 2002-12-20 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-02

CONDITIONS: Acute Traumatic Stress Disorders; Post-Traumatic Stress Disorders
Keywords: Acute Stress Disorder; PTSD; Treatment; SSRI; Startle; Psychophysiology; Trauma; Anxiety; Emotion
MeSH Terms: conditions — Stress Disorders, Traumatic, Acute; Stress Disorders, Post-Traumatic; Wounds and Injuries; Anxiety Disorders | interventions — Sertraline

INTERVENTIONS:
Drug: sertraline

SUMMARY:
The purpose of this study is to examine the short-term consequences of trauma and to determine the effectiveness of the drug sertraline in preventing and treating post-traumatic stress disorder (PTSD) and acute stress disorder (ASD) symptoms.

ASD and PTSD are common consequences of exposure to traumatic events. Despite growing evidence of neurobiological dysfunction in ASD and PTSD, the origin of these disorders is still unknown. This study will attempt to identify psychophysiological markers of ASD and find an effective treatment for its symptoms.

Victims of serious motor vehicle collisions will be evaluated with clinical assessments and standardized questionnaires within 2 weeks after the accident. Symptoms of exaggerated startle, emotional reactivity to trauma-related and trauma-unrelated cues, and cerebellum functioning will be evaluated. Participants will be randomized to receive either sertraline or placebo (an inactive sugar pill) for 8 weeks. Psychometric testing and psychological evaluations will be conducted 4, 10, and 14 weeks after the accident and after a 2-week taper of the study medication.

DETAILED DESCRIPTION:
Acute stress disorder (ASD) and posttraumatic stress disorder (PTSD) are common consequences of exposure to traumatic events. Despite growing evidence of neurobiological dysfunction in ASD and PTSD, the pathogenesis of these disorders is still unknown. Drs. Osuch and Ursano (Uniformed Services University of the Health Sciences) have received support to conduct a 14-week study that will investigate the efficacy of the serotonergic medication sertraline (Zoloft) in the treatment and prevention of posttraumatic psychiatric sequelae in ASD victims. The present project is an amendment to Drs. Osuch and Ursano's study. It will attempt to identify early psychological and neurobiological abnormalities in ASD. More specifically, the present project will examine to what extent sensitization and conditioning processes, as well as emotional dysregulation, contribute to ASD. We also propose to investigate the potential association between cerebellum dysfunction and peritraumatic dissociations. To accomplish this goal, a series of three experiments will be implemented to investigate: 1) the symptom of exaggerated startle; 2) emotional reactivity to trauma-related and trauma-unrelated cues; and 3) cerebellum functioning using eyeblink conditioning. This study will inform on the short-term consequences of trauma, will help identify potential psychophysiological markers of ASD that emerge following trauma, and will examine the effects of an SSRI on preventing trauma-related neurobiological deficits.

We specifically propose to:

1. Characterize psychophysiological responses in ASD victims shortly after trauma;
2. Assess the effect of sertraline treatment on these psychophysiological responses.

To accomplish aim 1, non-treated ASD victims will be compared to two control groups, a non-ASD trauma group and a non-trauma healthy group. The two control groups will be used to disentangle the effect of trauma from the effect of acute stress disorder. To accomplish aim 2, the ASD sertraline group will be compared to the ASD placebo group following treatment.

Forty victims of serious motor vehicle collision (MVC) with ASD will be recruited from a community hospital emergency room and evaluated with clinical assessments, and standardized questionnaires within 2 weeks after the MVC. The subjects will then be randomized to either sertraline or placebo for 8 weeks duration. Psychometric testing and psychological evaluations will be conducted at 4, 10 weeks post-MVC, and after a 2-week taper of the medication and 2 more weeks (14 weeks post-MVC).

We hypothesize that ASD patients will show:

An enhancement or sensitization of baseline startle;

An increase in autonomic arousal and in startle amplitude to trauma-related cues;

A delayed eyeblink conditioning;

Normalization of these deficits after sertraline treatment.

This preliminary study is expected to lay the groundwork for a larger study of the early impact of traumatic events on psychophysiological and psychological processes. In the long-term, we expect to 1) better characterize the onset of symptoms and their evolution over time following trauma, 2) identify psychophysiological markers for PTSD, 3) identify ASD victims at-risk for PTSD, and 4) improve our ability to prevent the development of chronic psychopathology following trauma.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects will be above seventh grade education level aged 18-65 years old and free of current or past psychopathology and organic central nervous system disorders that may interfere with the tests.

EXCLUSION CRITERIA:

Ongoing medical illness that may interfere with the tests; psychiatric or neurological disorder (including seizure); Past or current substance abuse; Current psychotropic medication; current medication that may interfere with the tests; Impaired hearing; major uncorrected visual impairment, or migraine headache.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2002-12; Study Completion 2004-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Harvey AG, Bryant RA. The relationship between acute stress disorder and posttraumatic stress disorder: a prospective evaluation of motor vehicle accident survivors. J Consult Clin Psychol. 1998 Jun;66(3):507-12. doi: 10.1037//0022-006x.66.3.507. PMID 9642889
- [Background] Harvey AG, Bryant RA. The relationship between acute stress disorder and posttraumatic stress disorder: a 2-year prospective evaluation. J Consult Clin Psychol. 1999 Dec;67(6):985-8. doi: 10.1037//0022-006x.67.6.985. PMID 10596520
- [Background] Blanchard EB, Hickling EJ, Taylor AE, Loos W. Psychiatric morbidity associated with motor vehicle accidents. J Nerv Ment Dis. 1995 Aug;183(8):495-504. doi: 10.1097/00005053-199508000-00001. PMID 7643060